CLINICAL TRIAL: NCT02139995
Title: West-China Transfusion Score for Critically-ill Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yiyun Deng, ICU, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ethics-42
Record Dates: First submitted 2014-05-11; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Transfusion Related Complication; Critical Illness
Keywords: transfusion; trigger; critically-ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transfusion trigger based on WCTS-CP (Experimental): Determination of whether a patient need red blood cells transfusion or which hemoglobin level should be maintained is based on WCTS-CP
  Interventions: Behavioral: RBC transfusion based on different protocols
- Transfusion trigger based on experience (Active Comparator): Determination of whether a patient need red blood cell transfusion or which hemoglobin level should be maintained is base on the physician's experience
  Interventions: Behavioral: RBC transfusion based on different protocols

INTERVENTIONS:
Behavioral: RBC transfusion based on different protocols — transfusion trigger for experimental group is the WCTS-CP；for active comparator is the physician's experience

SUMMARY:
Guidelines for blood transfusion have been issued for years. According to these guidelines, red blood cells (RBCs) transfusion should be given when the hemoglobin level is less than 6g/dL or 7g/dL and is unnecessary when the level is more than 10g/dL. However, in all the guidelines, the determination of whether RBCs should be administered when the hemoglobin level is in the range of 6~10g/dL is based on the judgment from doctors. Index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL is necessary and important in clinical practice.

Based on the aim of blood transfusion that maintain the balance of oxygen supply and oxygen consumption, the investigators hypothesize that index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL could be calculated by parameters including infusion rate of inotropic drugs for maintaining normal cardiac output, fraction of inspired oxygen, core temperature, and torlerance to anemia. To verify this hypothesis, the investigators present West China Transfusion Score for Critically-ill Patients(WCTS-CP) for the trigger of transfusion according to the patient's history and monitoring parameters, and the investigators design a randomized controlled clinical trial to test this score.

DETAILED DESCRIPTION:
Anemia is a common phenomenon in critically ill patients, and blood transfusion may provide guarantee for oxygen delivery. On the other hand, blood transfusion is associated with many risks including hemolytic and nonhemolytic reactions, transfusion related acute lung injury (TRALI), and others. Besides, blood is insufficient worldwide. How to eliminate allogeneic blood transfusion is an important part in clinical practice.

Guidelines for blood transfusion have been issued for years. According to these guidelines, red blood cells (RBCs) transfusion should be given when the hemoglobin level is less than 6g/dL or 7g/dL and is unnecessary when the level is more than 10g/dL. However, in all the guidelines, the determination of whether RBCs should be administered when the hemoglobin level is in the range of 6~10g/dL is based on the judgment from specific doctors. Index of transfusion trigger for critically ill patients with hemoglobin level between 6g/dL and 10g/dL is necessary and important in clinical practice.

Based on the aim of blood transfusion that maintain the balance of oxygen supply and oxygen consumption, the investigators hypothesize that index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL could be calculated by parameters including infusion rate of inotropic drugs for maintaining normal cardiac output, fraction of inspired oxygen for maintaining saturation of oxygen≧95%, core temperature, and torlerance to anemia.

The investigators set down the West China Transfusion Score for Critically-ill Patients(WCTS-CP) ，the initial score is 6. If a patient's cardiac output is normal without infusion of inotropic drugs, the heartbeat less than 100 per minute，his saturation of oxygen could be maintained more than 95%, his core temperature is less than 38℃, and he has no history of ischemic cardiovascular disease , and he is below 55 of age，his score is 6.

If a patient has one or more problems, his score should be added 1 point for each problem.

The initial WCTS-CP score is 6, and the patient's score is calculated by the sum of each item.

Score 6：The transfusion trigger is 6g/dL, and the the patient's Hemoglobin level should be maintained not less than 6g/dL.

Score 7：The transfusion trigger is 7g/dL, and the the patient's Hemoglobin level should be maintained not less than 7g/dL.

Score 8：The transfusion trigger is 8g/dL, and the the patient's Hemoglobin level should be maintained not less than 8g/dL.

Score 9：The transfusion trigger is 9g/dL, and the the patient's Hemoglobin level should be maintained not less than 9g/dL.

Score 10 or >10：The transfusion trigger is 10g/dL, and the the patient's Hemoglobin level should be maintained not less than 10g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Height of usual place of residence less than 2,500 metres above sea level
* Hemoglobin level possibly less than 10g/dL

Exclusion Criteria:

* Pregnant women
* Age less than 18
* Serious blood system diseases
* Dysfunction of hemoglobin
* Tumor metastasis
* Psychopathy
* Refuse to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of death and serious complications | 28 days

SECONDARY OUTCOMES:
Transfusion rate and transfusion volume of red blood cells | 28 days
ventilator-free days in 28 days | 28 days
  The time that patients do not need ventilaton support
length of stay in ICU or in hospital | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, M.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China